CLINICAL TRIAL: NCT05084521
Title: Interest of Famotidine in Reducing Endothelial Expression of P-selectin in Children With Sickle Cell Disease: Pilot Study, Single-center, Prospective, Non-comparative.
Brief Title: Interest of Famotidine in Children With Sickle Cell Disease
Acronym: FAMODREP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: INSERM U 1163 - Laboratory of molecular mechanisms of hematologic disorders and therapeutic implications, Paris (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP201133; 2021-001351-13 (EudraCT Number)
Record Dates: First submitted 2021-10-15; First posted 2021-10-19 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Sickle Cell Disease
Keywords: Sickle cell disease; Famotidine; Histamine; P-selectin; Vaso-occlusive crisis
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises | interventions — Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Famotidine (Experimental): Suspension of famotidine, 0.5 mg/kg/12h (with a maximum dose of 80 mg/day, regardless of the patient's weight) during 29 days.
  Interventions: Drug: Famotidine 400 mg/50 mL

INTERVENTIONS:
Drug: Famotidine 400 mg/50 mL — Administration of a suspension of famotidine, 0.5 mg/kg/12h (with a maximum dose of 80 mg/day, regardless of the patient's weight) during 29 days.

SUMMARY:
The purpose of this study is to determine whether oral famotidine, a histamine type 2 receptor antagonist already widely used with very few side effects in other indications in children, is effective in reducing endothelial expression of P-selectin in children with sickle cell disease (SCD).

This pilot study will constitute the essential prerequisite for a randomized clinical trial comparing the efficacy of famotidine with that of placebo in the prevention of vaso-occlusive crises in SCD patients.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is a frequent and severe hemoglobinopathy, considered the first monogenic disease in the world. It is responsible for chronic hemolytic anemia, painful vaso-occlusive crises secondary to obstruction of the microcirculation by sickled red blood cells adhering to the vascular endothelium, and progressive organ damage secondary to ischemia/reperfusion phenomena.

Although the molecular bases are well known, the pathophysiology is still incompletely understood and therapeutic options remain limited. We have recently demonstrated an increase in plasma histamine levels (associated with mast cell activation) in SCD patients, particularly ≤ 18 years of age, at baseline and even more markedly during vaso-occlusive crises (Allali, Br J Haematol 2019). In vitro, an increase in the adhesion of red blood cells of SCD patients to human endothelial cells after stimulation with histamine has been described, via an increased expression of the adhesion molecule P-selectin. Abolition of this effect in the presence of famotidine, a histamine type 2 (H2) receptor antagonist, suggests that histamine is responsible for an increased adhesion mediated by P-selectin via stimulation of the H2 receptors. Therefore, our hypothesis is that long-term use of oral antihistamine therapy with famotidine may prevent vaso-occlusion by decreasing P-selectin expression by endothelial cells.

The main objective of the study is to assess the effect of famotidine on P-selectin expression after 29 days of oral treatment.

The secondary objectives are:

* to assess the effect of famotidine on the expression of other endothelial activation markers after 29 days of treatment;
* to assess the effect of famotidine on biomarkers of hemolysis and inflammation after 29 days of treatment;
* to assess the adverse effects of famotidine in a pediatric population suffering from sickle cell disease.

The experimental design will be a monocentric, prospective, non-comparative, pilot cohort study. The population studied will be that of children aged 1 to 17 years and 10 months, followed at the Necker-Enfants malades hospital for SS or Sβ0 SCD and having presented at least one vaso-occlusive crisis during the year prior to inclusion. All the children included will be treated for 29 days with famotidine in oral suspension, at a dosage of 0.5 mg/kg/12h (with a maximum dose of 80 mg/day, regardless of the patient's weight). Patient recruitment will take place in the General Pediatrics and Infectious Diseases department/SCD Center of the Necker-Enfants malades Hospital in consultation or during hospitalization. The selection visit will take place 3 months before the inclusion visit and the research itself will comprise 3 visits (D0, D29 and D36/End of study).

Treatment will be started on D1, in the morning.

During the inclusion visit will be carried out:

* verification of inclusion and non-inclusion criteria;
* obtention of the consent of the 2 parents/legal representative(s) and of the child;
* a complete clinical examination;
* a biological assessment including a plasma assay of P-selectin, E-selectin, VCAM-1 and ICAM-1 by ELISA technique, in the research laboratory of Prof. Olivier Hermine (Imagine Institute), and examinations carried out as part of the usual follow-up for SCD children in the routine laboratories of the Necker-Enfants malades hospital: complete blood count, reticulocyte count, C-reactive protein, serum urea, creatinine, and electrolytes, aspartate and alanine aminotransferase, total and direct bilirubin, gamma-glutamyl transferase, lactate dehydrogenase, and hemoglobin S/F. A plasma histamine assay will also be carried out in the immunology laboratory of the Bichat-Claude Bernard hospital.

During the follow-up visit at D29, will be carried out:

* a questioning on possible symptoms (pain, headache, feeling of dizziness, transit disorders, etc.) and on adherence to treatment since the inclusion visit (using a logbook for monitoring tolerance and compliance);
* a complete clinical examination identical to that of the inclusion visit;
* a biological assessment identical to that carried out during the inclusion visit (except for HbS/F assay which will not be performed).

Famotidine treatment will be discontinued at the end of this research visit. A phone call is scheduled 7 days after stopping treatment to monitor the occurrence of adverse events (i.e. on D36) and will correspond to the end of the research.

The various visits will be carried out by the principal investigator or by his collaborators (registered pediatricians and trained in research from the General Pediatrics and Infectious Diseases Department/SCD Center).

The number of patients to be included will be 30, or 2 to 3 patients/month for 12 months. The total duration of the research will be 13 months and 1 week:

* selection period: 3 months
* duration of inclusion: 12 months
* duration of participation (treatment + follow-up): 29 + 7 days
* duration of treatment: 29 days (between 26 and 29 days)

This study of the effect of famotidine on the expression of P-selectin in children with SCD will constitute the essential prerequisite for the performance of a randomized clinical trial comparing the efficacy of famotidine with that of a placebo in the prevention of vaso-occlusive crises.

Oral antihistamine treatment with famotidine, which is already widely used with very few side effects in other indications in children, may constitute an inexpensive, original and innovative therapeutic approach in SCD.

ELIGIBILITY:
Inclusion Criteria:

* child or adolescent aged 1 year to 17 years and 10 months, followed at the Necker-Enfants malades Hospital for a SS or Sβ0 SCD;
* having at least one vaso-occlusive crisis in the year prior to inclusion;
* for young girl of childbearing age (≥ 15 years old), a negative pregnancy test;
* signed informed consent of the 2 parents or legal representative(s) and of the child of expressive age or the adolescent;
* beneficiary of social security coverage or entitled (excluding AME)

Exclusion Criteria:

* treatment with crizanlizumab (anti-P-selectin antibody);
* treatment with atazanavir/ritonavir in combination with tenofovir;
* known hypersensitivity to famotidine or to other histamine type 2 (H2) receptor antagonists;
* cardiovascular history such as: arrhythmia, AVB (atrioventricular block), QT prolongation;
* renal failure characterized by creatinine clearance <60 mL/min;
* hepatic cytolysis (ALT ≥ 3N);
* neutropenia (<1 G/L), thrombocytopenia (<80 G/L), reticulopenia (<80 G/L);
* predictable poor adherence to treatment;
* pregnancy or breastfeeding;
* participation in another interventional research involving the human person;
* planned bone marrow transplant or gene therapy within one month of inclusion.

Within 3 months prior to inclusion:

* red blood cell transfusion;
* introduction of hydroxyurea or modification of hydroxyurea doses;
* introduction of L-glutamine or modification of L-glutamine doses;
* introduction of voxelotor or modification of voxelotor doses;
* taking oral or IV corticosteroids or any other immunomodulatory treatment;
* taking an antihistamine treatment

In the month preceding inclusion:

* occurrence of a vaso-occlusive crisis, acute chest syndrome or any vaso-occlusive phenomenon (acute splenic sequestration, priapism, stroke, occlusion of the central retinal artery, papillary necrosis);
* occurrence of fever (≥ 38°C) or any infectious episode, febrile or not, suspected or confirmed, of a viral, bacterial, fungal or parasitic nature ;
* occurrence of an acute hemolytic episode (increase in jaundice and pallor, decrease in hemoglobin level of ≥ 1 g/dL compared to baseline hemoglobin, increase in LDH and/or AST and/or free bilirubin deemed significant by the child's referring physician).

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Difference in plasma concentration of soluble P-selectin | 29 days
  Measurement by ELISA technique before and after 29 days of treatment

SECONDARY OUTCOMES:
Difference in plasma concentration of soluble adhesion molecule: E-selectin | 29 days
  Measurement by ELISA technique before and after 29 days of treatment
Difference in plasma concentration of soluble adhesion molecule: VCAM-1 | 29 days
  Measurement by ELISA technique before and after 29 days of treatment
Difference in plasma concentration of soluble adhesion molecule: ICAM-1 | 29 days
  Measurement by ELISA technique before and after 29 days of treatment
Differences in blood values: hemoglobin, reticulocytes, AST, free bilirubin, LDH, and CRP | 29 days
  Dosage on D0 and D29
Occurrence of serious or non-serious adverse event(s) | 36 days
Occurrence of vaso-occlusive crisis | 36 days

CONTACTS AND LOCATIONS:
Overall Officials: Slimane ALLALI, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Olivier HERMINE, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Necker - Enfants malades Hospital; Department of Pediatrics and Infectious Diseases, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Allali S, Marquant F, Rignault-Bricard R, Taylor M, Brice J, de Montalembert M, Maciel TT, Elie C, Hermine O. Oral famotidine reduces the plasma level of soluble P-selectin in children with sickle cell disease. Br J Haematol. 2024 Jan;204(1):346-351. doi: 10.1111/bjh.19111. Epub 2023 Sep 18. PMID 37722599